CLINICAL TRIAL: NCT06862115
Title: The Effect of Discontinuation of Renin Angiotensin System Inhibitors on the Perioperative Myocardial Injury in Adult Patients Undergoing Colorectal Cancer Surgery: a Randomized Controlled Non Inferiority Study.
Brief Title: The Effect of Discontinuation of Renin Angiotensin System Inhibitors on the Perioperative Myocardial Injury in Adult Patients Undergoing Colorectal Cancer Surgery
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MS-525-2024
Record Dates: First submitted 2025-03-01; First posted 2025-03-06 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Myocardium; Injury; Perioperative/Postoperative Complications; Angiotensin-Converting-Enzyme Inhibitor
MeSH Terms: conditions — Wounds and Injuries; Postoperative Complications

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Trial participants and staff will not be blinded to treatment group allocation however, all investigators will be blinded to the primary outcome measure (myocardial injury).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stop RAS (Experimental): When the ACE-I and/or ARB duration of action is ≥24 hours, the drug will be stopped 48 hours prior to surgery. All other ACE-I and/or ARB will be stopped 24 hours before surgery.
  Interventions: Drug: ACE-I and/or ARB antihypertensive treatment
- continue RAS (Active Comparator): ACE-I and ARBs will be continued till morning of surgery
  Interventions: Drug: ACE-I and/or ARB antihypertensive treatment

INTERVENTIONS:
Drug: ACE-I and/or ARB antihypertensive treatment — When the ACE-I and/or ARB duration of action is ≥24 hours, the drug will be stopped 48 hours prior to surgery. All other ACE-I and/or ARB will be stopped 24 hours before surgery.

SUMMARY:
The aim of this study is to estimate the effect of discontinuation of RAS inhibitors on myocardial injury in cancer patients undergoing major abdominal surgeries.

DETAILED DESCRIPTION:
This is a prospective, open-label, randomized controlled non inferiority trial. Participants will be assigned randomly in a 1:1 manner whether to stop or continue RAS inhibitors. Randomization will be performed using an online program (www.randomizer.com).

Trial participants and staff will not be blinded to treatment group allocation however, all investigators will be blinded to the primary outcome measure (myocardial injury).

After randomization during the preoperative visit, participants will be instructed to stop or continue their ACE-I and/or ARB according to their allocated group. ACE-I and/or ARB will be continued or discontinued as per treatment group allocation and this will continue until 24 hours after the end of surgery. Since ACE-I and ARB have different durations of action, participants will receive drug-specific instructions as to when to stop. When the ACE-I and/or ARB duration of action is ≥24 hours, the drug will be stopped 48 hours prior to surgery. All other ACE-I and/or ARB will be stopped 24 hours before surgery. Renin-angiotensin system inhibitors will be restarted after surgery on the morning of post-operative day one if systolic blood pressure was >120 mmHg in the previous 12 hours.

The anesthetic induction, intraoperative and postoperative management will be managed according to the local policy of the NCI by expert anesthesiologists who will be blinded to the patients' groups.

Troponin-I will be measured at 9 a.m. on the day before surgery and at 9 a.m. on postoperative day one and day two. Myocardial injury will be defined as: (Troponin-I an increase by 0.015 is considered positive, if the baseline is <0.05 A. If the baseline is higher than 0.05, an increase by 0.005 is considered positive).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Both sexes
* ASA 2-3
* Chronic hypertensive patients (> 3 months before surgery) controlled on ACEIs or ARBs or combination therapy containing one of the RAS inhibitors.
* Scheduled for major abdominal cancer surgery (surgery with an expected duration of > 2 h from the surgical incision and a postoperative hospital stay of least three days).

Exclusion Criteria:

* Patient refusal.
* Recent myocardial infarction (within 3 months).
* Any condition, which in the opinion of the treating clinician, would result in the patient being harmed by the cessation of the ACE-I and/or ARB therapy.
* Emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the incidence of myocardial injury 48 hours after surgery | 48 hours
  defined as: (Troponin-I If the baseline is <0.05 And increase by 0.015 is considered positive
  If the baseline is higher than 0.05, an increase by 0.005 is considered positive

SECONDARY OUTCOMES:
Highest level of Troponin-I measured within 48 hours of surgery. | 48 hours
  Highest level of Troponin-T measured within 48 hours of surgery.
Incidence of perioperative hypotension | 48 hours
  Incidence of perioperative hypotension (MAP<20% of baseline measure recorded night before surgery) until 48 hours after surgery.
Incidence of severe hypotension | 48 hours
  Incidence of severe hypotension (MAP < 60 mmHg requiring any vasopressor) until 48 hours after surgery.
Incidence of perioperative severe hypertension | 48 hours
  Incidence of perioperative severe hypertension (BP>180/100mmHg) until 48 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided